CLINICAL TRIAL: NCT07325877
Title: Supra-papillary Versus Trans-papillary Biliary Stenting in Malignant Peri-hilar Stenosis (SupraBilS): a Randomized Controlled Trial
Brief Title: Supra-papillary Versus Trans-papillary Biliary Stenting in Malignant Peri-hilar Stenosis
Acronym: SupraBilS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Andrea Ruzzenente, Professor, Azienda Ospedaliera Universitaria Integrata Verona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ID0001; ID0001 (Other: Integrated University Hospital Verona)
Record Dates: First submitted 2025-12-16; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Biliary Disease Tract; Biliary Stenosis; Biliary Stents
Keywords: ERCP; Malignant Biliary Stenosis; Supra-papillary; Trans-Papillary
MeSH Terms: conditions — Biliary Tract Diseases | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Intervention Model Description: This is a single-blinded randomized controlled trial comparing two techniques used for the same procedure (ERCP and biliary stenting, suprapapillary vs transpapillary placement).
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suprapapillary (Experimental): ERCP for malignant stenosis of bile duct with suprapapillary stents positioning (experimental)
  Interventions: Procedure: ERCP with suprapapillary stent placement
- Trans Papillary (Active Comparator): ERCP for malignant stenosis of bile duct with transpapillary stents positioning (Standard of care).
  Interventions: Procedure: ERCP with transpapillary stent placement

INTERVENTIONS:
Procedure: ERCP with suprapapillary stent placement — ERCP with no sphincterotomy and placement of plastic stents above the papilla of Vater.
  Arms: Suprapapillary
Procedure: ERCP with transpapillary stent placement — Standard ERCP with or without sphincterotomy with trans papillary stent placement
  Arms: Trans Papillary

SUMMARY:
This is a randomized controlled trial comparing patients with obstructive jaundice due to malignancies of the perihilar area of bile ducts and undergoing both preoperative and palliative biliary drainage. The comparison will focus on the technique:, on the one hand, an arm of patients undergoing standard-of-care ERCP with trans-papillary plastic protesis placement, and on the other hand, an experimental arm of patients undergoing suprapapillary plastic protesis placement with no sphincterotomy. The primary objective will be to compare the time-to-stent dysfunction in the two groups; secondary objectives will include a comparison of the safety, technical, and clinical success of the procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Radiological/ biochemical/pathological diagnosis of malignant OJ.
2. Stenosis maximum extent may be 2 cm after biliary confluence.
3. Documented obstructive jaundice (serum bilirubin > 3 mg/dL).
4. Indication for biliary drainage (preoperative or palliative).
5. Age ≥ 18 years.
6. Signed informed consent.

Exclusion Criteria:

1. Contraindications to endoscopic approach (duodenal stenosis, surgically altered anatomy).
2. Previous sphincterotomy or drainage.
3. Involvement of the papilla of Vater by the tumour.
4. Uncontrolled coagulopathy (INR > 1.5 uncorrectable or <50.000 PLTs).
5. Ongoing uncontrolled cholangitis as defined according to the Tokyo 2018 Guidelines, or systemic sepsis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Time-to-Stent disfunction | From index procedure to a minimum of one year of follow up.
  In days, calculated from the index procedure. Stent(s) dysfunction, which includes occlusion or migration of the stent(s) and tumour ingrowth/overgrowth, is defined as the presence of at least two of the following three criteria:
  1. New dilation of the biliary tree on imaging:
  2. Bilirubin level above 2 mg/dL (34.2 mmol/L) with a new increase ≥ 1 mg/dL compared with the value after initial clinical success, or elevation of alkaline phosphatase and/or g-glutamyl transferase greater than 2 times the upper normal limit with a new elevation of 30 U/L
  3. Cholangitis, characterized by fever along with leucocytosis (> 10,000/mL) or C-reactive protein levels above 20 mg/dL.

SECONDARY OUTCOMES:
Safety of the procedure | From the index procedure within 14 days.
  The incidence of Adverse events and severe adverse events will be compared. Adverse events (AEs) (timepoint 14 days) are defined according to the ASGE lexicon and graded according to the Adverse Events in GI endoscopy (AGREE) classification that classifies AEs in 5 grades from Grade I, any deviation from standard postprocedural course without need for pharmacological or interventional treatment, to Grade V, death of the patient. Sub-group analysis will be performed for procedure-related AEs. Severe adverse events are defined as AGREE≥3.
Technical success | At the moment of index procedure.
  Defined as the placement of the stent(s) in the desired position (timepoint 0)
Clinical Success | Between 14 and 30 days from the index procedure.
  Defined as the reduction of bilirubin level ≥50% or at a level <2 mg/dL (34.2 mmol/L).

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Ruzzenente, Professor, Principal Investigator — Integrated University Hospital Verona; Stefano Francesco Crinò, Consultant, Study Director — Integrated University Hospital Verona; Edoardo Poletto, PhD Candidate, Consultant, Study Chair — Integrated university Hospital Verona; Maria Cristina Conti Bellocchi, Consultant, Study Chair — Integrated University Hospital Verona

IPD SHARING:
Plan to Share IPD: Undecided
Question asked to the ethics committee, decision is still pending.

REFERENCES:
- [Background] Naitoh I, Inoue T. Optimal endoscopic drainage strategy for unresectable malignant hilar biliary obstruction. Clin Endosc. 2023 Mar;56(2):135-142. doi: 10.5946/ce.2022.150. Epub 2023 Jan 5. PMID 36600654
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660
- [Background] Kiriyama S, Kozaka K, Takada T, Strasberg SM, Pitt HA, Gabata T, Hata J, Liau KH, Miura F, Horiguchi A, Liu KH, Su CH, Wada K, Jagannath P, Itoi T, Gouma DJ, Mori Y, Mukai S, Gimenez ME, Huang WS, Kim MH, Okamoto K, Belli G, Dervenis C, Chan ACW, Lau WY, Endo I, Gomi H, Yoshida M, Mayumi T, Baron TH, de Santibanes E, Teoh AYB, Hwang TL, Ker CG, Chen MF, Han HS, Yoon YS, Choi IS, Yoon DS, Higuchi R, Kitano S, Inomata M, Deziel DJ, Jonas E, Hirata K, Sumiyama Y, Inui K, Yamamoto M. Tokyo Guidelines 2018: diagnostic criteria and severity grading of acute cholangitis (with videos). J Hepatobiliary Pancreat Sci. 2018 Jan;25(1):17-30. doi: 10.1002/jhbp.512. Epub 2018 Jan 5. PMID 29032610
- [Background] Nass KJ, Zwager LW, van der Vlugt M, Dekker E, Bossuyt PMM, Ravindran S, Thomas-Gibson S, Fockens P. Novel classification for adverse events in GI endoscopy: the AGREE classification. Gastrointest Endosc. 2022 Jun;95(6):1078-1085.e8. doi: 10.1016/j.gie.2021.11.038. Epub 2021 Dec 8. PMID 34890695
- [Background] Cotton PB, Eisen GM, Aabakken L, Baron TH, Hutter MM, Jacobson BC, Mergener K, Nemcek A Jr, Petersen BT, Petrini JL, Pike IM, Rabeneck L, Romagnuolo J, Vargo JJ. A lexicon for endoscopic adverse events: report of an ASGE workshop. Gastrointest Endosc. 2010 Mar;71(3):446-54. doi: 10.1016/j.gie.2009.10.027. No abstract available. PMID 20189503
- [Background] Kovacs N, Pecsi D, Sipos Z, Farkas N, Foldi M, Hegyi P, Bajor J, Eross B, Marta K, Miko A, Rakonczay Z Jr, Sarlos P, Abraham S, Vincze A. Suprapapillary Biliary Stents Have Longer Patency Times than Transpapillary Stents-A Systematic Review and Meta-Analysis. J Clin Med. 2023 Jan 23;12(3):898. doi: 10.3390/jcm12030898. PMID 36769545
- [Background] Okamoto T, Fujioka S, Yanagisawa S, Yanaga K, Kakutani H, Tajiri H, Urashima M. Placement of a metallic stent across the main duodenal papilla may predispose to cholangitis. Gastrointest Endosc. 2006 May;63(6):792-6. doi: 10.1016/j.gie.2005.05.015. PMID 16650540
- [Background] Keulen AV, Gaspersz MP, van Vugt JLA, Roos E, Olthof PB, Coelen RJS, Bruno MJ, van Driel LMJW, Voermans RP, van Eijck CHJ, van Hooft JE, van Lienden KP, de Jonge J, Polak WG, Poley JW, Pek CJ, Moelker A, Willemssen FEJA, van Gulik TM, Erdmann JI, Hol L, IJzermans JNM, Buttner S, Koerkamp BG. Success, complication, and mortality rates of initial biliary drainage in patients with unresectable perihilar cholangiocarcinoma. Surgery. 2022 Dec;172(6):1606-1613. doi: 10.1016/j.surg.2022.06.028. Epub 2022 Aug 18. PMID 35989132
- [Background] Ipek S, Alper E, Cekic C, Cerrah S, Arabul M, Aslan F, Unsal B. Evaluation of the effectiveness of endoscopic retrograde cholangiopancreatography in patients with perihilar cholangiocarcinoma and its effect on development of cholangitis. Gastroenterol Res Pract. 2014;2014:508286. doi: 10.1155/2014/508286. Epub 2014 May 27. PMID 24982670
- [Background] Vogel A, Bridgewater J, Edeline J, Kelley RK, Klumpen HJ, Malka D, Primrose JN, Rimassa L, Stenzinger A, Valle JW, Ducreux M; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Biliary tract cancer: ESMO Clinical Practice Guideline for diagnosis, treatment and follow-up. Ann Oncol. 2023 Feb;34(2):127-140. doi: 10.1016/j.annonc.2022.10.506. Epub 2022 Nov 10. No abstract available. PMID 36372281
- [Background] Qumseya BJ, Jamil LH, Elmunzer BJ, Riaz A, Ceppa EP, Thosani NC, Buxbaum JL, Storm AC, Sawhney MS, Pawa S, Naveed M, Lee JK, Law JK, Kwon RS, Jue TL, Fujii-Lau LL, Fishman DS, Calderwood AH, Amateau SK, Al-Haddad M, Wani S. ASGE guideline on the role of endoscopy in the management of malignant hilar obstruction. Gastrointest Endosc. 2021 Aug;94(2):222-234.e22. doi: 10.1016/j.gie.2020.12.035. Epub 2021 May 20. PMID 34023067
- [Background] Boulay BR, Birg A. Malignant biliary obstruction: From palliation to treatment. World J Gastrointest Oncol. 2016 Jun 15;8(6):498-508. doi: 10.4251/wjgo.v8.i6.498. PMID 27326319
- [Background] Hameed A, Pang T, Chiou J, Pleass H, Lam V, Hollands M, Johnston E, Richardson A, Yuen L. Percutaneous vs. endoscopic pre-operative biliary drainage in hilar cholangiocarcinoma - a systematic review and meta-analysis. HPB (Oxford). 2016 May;18(5):400-10. doi: 10.1016/j.hpb.2016.03.002. Epub 2016 Apr 4. PMID 27154803
- [Background] Pavlidis ET, Pavlidis TE. Pathophysiological consequences of obstructive jaundice and perioperative management. Hepatobiliary Pancreat Dis Int. 2018 Feb;17(1):17-21. doi: 10.1016/j.hbpd.2018.01.008. Epub 2018 Jan 31. PMID 29428098
- [Background] Ruzzenente A, Alaimo L, Caputo M, Conci S, Campagnaro T, De Bellis M, Bagante F, Pedrazzani C, Guglielmi A. Infectious complications after surgery for perihilar cholangiocarcinoma: A single Western center experience. Surgery. 2022 Sep;172(3):813-820. doi: 10.1016/j.surg.2022.04.028. Epub 2022 May 24. PMID 35618490
- [Background] Valle JW, Kelley RK, Nervi B, Oh DY, Zhu AX. Biliary tract cancer. Lancet. 2021 Jan 30;397(10272):428-444. doi: 10.1016/S0140-6736(21)00153-7. PMID 33516341